CLINICAL TRIAL: NCT02512471
Title: The Minimum Effective Volume of Ropivacaine in Ultrasound-guided Supraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Fang Gang, Dr., Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-64-2
Record Dates: First submitted 2015-07-25; First posted 2015-07-31 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Supraclavicular Brachial Plexus Block
Keywords: minimum effective volume; ropivacaine; ultrasound-guided supraclavicular block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- middle aged group (Experimental): brachial plexus block with ropivacaine 0.275%, MEV90 for USG-SCB
  Interventions: Drug: Ropivacaine
- young group (Active Comparator): brachial plexus block with ropivacaine 0.325%, MEV90 for USG-SCB
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — brachial plexus block with ropivacaine 0.275%, MEV90 for USG-SCB (young group) brachial plexus block with ropivacaine 0.325%, MEV90 for USG-SCB (middle-aged group)
  Other Names: Naropin

SUMMARY:
The aim of this study is to determine the minimum effective volume of local anesthetic (ropivacaine 0.275% and 0.325%) required to produce an effective double-injection USG-SCB for surgical anesthesia in 90% of patients (MEV90) in young group (18-40 years) and in middle aged group (40-65 years) of patients scheduled for elective surgery of one upper limb distal to the shoulder.

DETAILED DESCRIPTION:
The study is based on biased coin design, and the volume of LA for the next patient is determined by the result of the last one. In the case of block failure, the volume will be increased by 2ml. Conversely, block success will result in either a reduction in volume by 2ml (probability 11%) or no change in volume (probability 89%). A blinded assistant will assess sensory and motor blockade in each nerve territory ( the median, radial, ulnar and musculocutaneous nerves) at 10-min intervals up to 30 min after completion of the block. Finally, MEV90 is calculated by isotonic regression.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years
2. ASA 1-3
3. body mass index between 18 and 35kg/m2

Exclusion Criteria:

1. inability to consent to the study
2. pregnancy
3. allergy to local anesthetics
4. preexisting neuropathy or coagulopathy
5. prior surgery in the supraclavicular region

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The Minimum Effective Volume of Ropivacaine in Ultrasound-guided Supraclavicular Block | up to 6 months
  The Minimum Effective Volume (MEV) of Ropivacaine in Ultrasound-guided Supraclavicular Block is based on 55 measurements in 55 patients (secondary outcome measure: block success). MEV is determined by biased coin design method when all patients have been tested in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ailin Luo, MD.,PhD, Study Chair — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China